CLINICAL TRIAL: NCT06919562
Title: OPtimal stEnt Deployment stRategy oF Contemporary sTents - Registry to Evaluate Percutaneous Coronary Intervention Using Bioresorbable Scaffolds With Thinner-strut Construction and Guidance by intracOronary Imaging to REduce Scaffold Failure
Acronym: PERFECTRESTORE
Status: Not yet recruiting | Type: Observational
Sponsor: Albert Schweitzer Ziekenhuis, Netherlands (Other)
Collaborators: Meril Life Sciences Pvt. Ltd. (Industry); Angiocare BV, Netherlands (Unknown); Salveo Medical BV, Netherlands (Unknown)
Responsible Party: Principal Investigator, Jin M. Cheng, MD, PhD, Albert Schweitzer Ziekenhuis, Netherlands
Other Study IDs: PERFECT RESTORE; NL-009177 (Other: CCMO)
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Coronary Arterial Disease (CAD); Percutaneous Coronary Intervention (PCI)
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Percutaneous coronary intervention with protocolized implantation of a second generation thin-strut bioresorbable scaffold guided by intracoronary imaging — Percutaneous coronary intervention (PCI) with implantation of the MeRes100 thin-strut BRS with protocolized PSP (predilatation, sizing, postdilatation) method and intracoronary imaging guidance.

SUMMARY:
Implantation of a metallic drug-eluting stent (DES) is currently the gold standard in percutaneous coronary intervention (PCI). However, a DES has several limitations on the long-term, such as chronic local inflammation which may lead to in-stent restenosis, absence of physiological coronary vasomotion and vessel caging which makes future coronary artery bypass grafting (CABG) impossible. A bioresorbable scaffold (BRS) is designed to overcome these limitations. The first generation BRS was shown to be clinically inferior to DES due to a slightly higher rate of stent thrombosis. To overcome this problem, several scientific developments have been achieved in the past few years, such as thinner BRS strut construction and improved implantation technique by using PSP (predilatation, sizing, postdilatation) method and intracoronary imaging guidance with optical coherence tomography (OCT) or intravasculair ultrasound (IVUS). A PCI protocol that combines implantation of a second generation thin-strut BRS, mandatory PSP implantation method and mandatory intracoronary imaging-guidance has not yet been investigated. The aim of this study is to investigate feasibility of a new PCI protocol with implantation of the second generation Meres100 thin-strut BRS combined with a protocolized PSP implantation technique guided by intracoronary imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Stable coronary artery disease with one or more significant epicardial stenosis in native coronary arteries suitable for OCT or IVUS-guided PCI with BRS implantation.
2. Subject must be at least 18 years of age
3. Written consent to participate in the study

Exclusion Criteria:

1. Culprit lesions in the setting of acute coronary syndrome.
2. Lesions with severe calcification.
3. Lesions in a coronary artery with severe tortuosity.
4. Left main coronary artery lesions.
5. Bifurcation lesions.
6. Ostial lesions.
7. Lesions with a difference in proximal and distal reference diameter of >0.5 mm by visual judgement of the coronary angiogram by the treating operator.
8. Treatment of in-stent restenosis or stent thrombosis.
9. History of definite stent thrombosis.
10. Lesions in coronary artery bypass grafts.
11. Lesions not suitable for OCT or IVUS catheter delivery and imaging, e.g. due to tortuosity or distal localisation.
12. Creatinine Clearance ≤ 30 ml/min/1.73 m2 as calculated by MDRD formula for estimated GFR.
13. Contraindication to dual antiplatelet therapy with aspirin and a P2Y12 inhibitor or (if indicated) NOAC and P2Y12 inhibitor.
14. Planned non-deferrable major surgery after PCI.
15. Known comorbidity associated with a life expectancy <1 year.
16. Unable to understand and follow study-related instructions or unable to comply with study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with obstructive stable coronary artery disease
Sampling Method: Probability Sample
Enrollment: 117 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Technical success | End of procedure
  Percentage of technical success, defined as successful implantation of the BRS in the obstructive coronary lesion.
Angiographic success | End of procedure
  Percentage of angiographic success, defined as <10% residual stenosis and TIMI 3 flow.
Treatment protocol adherence | End of procedure
  Percentage of treatment protocol adherence, defined as full completion of all PSP and intracoronary imaging steps during implantation procedure.
Optimal scaffold result | End of procedure
  Percentage of optimal scaffold result on intracoronary imaging, defined as no major edge dissection, no major malexpansion and scaffold expansion >90%.
Additional optimization steps | End of procedure
  Percentage of additional optimization steps (including additional postdilatation, additional BRS implantation, bailout metallic DES implantation, additional intracoronary imaging) to achieve optimal scaffold result.
Target Lesion Failure | 1-year and 3-year post-procedure
  Estimate of target lesion failure (TLF), defined as the composite of cardiovascular death, target-vessel related myocardial infarction and clinically driven target lesion revascularization
Scaffold thrombosis | 1-year and 3-year post-procedure
  Estimate of scaffold thrombosis

SECONDARY OUTCOMES:
Minimal scaffold area | End of procedure
  Minimal scaffold area assessed with the final OCT or IVUS measurement
Scaffold malapposition | End of procedure
  Scaffold malapposition as percentage, defined as frequency of incompletely apposed struts (i.e. struts clearly separated from the vessel wall without any tissue behind the struts with a distance from the adjacent intima of ≥0.2 mm and not associated with any side branch) assessed with the final OCT or IVUS measurement.
Scaffold expansion | End of procedure
  Scaffold expansion as percentage, defined as scaffold area divided by the average of proximal and distal reference lumen areas, assessed with the final OCT or IVUS measurement.
Edge dissection | End of procedure
  Presence of edge dissection assessed with the final OCT or IVUS measurement.
Intra-scaffold plaque protrusion and thrombus | End of procedure
  Intra-scaffold plaque protrusion and thrombus, defined as any intraluminal mass protruding at least 0.2 mm within the luminal edge of a stent strut, assessed with the final OCT or IVUS measurement.

IPD SHARING:
Plan to Share IPD: Yes